CLINICAL TRIAL: NCT04704466
Title: Observational Study Evaluating the Impact of the Covid-19 Pandemic on the Management of Patients With Head and Neck Cancer in the Maxillofacial Surgery Department
Brief Title: Impact of Covid-19 Pandemic on Management of Head and Neck Cancers
Acronym: VADS-Covid
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0003
Record Dates: First submitted 2021-01-08; First posted 2021-01-11 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Head and Neck Cancer; Covid19; Patient Care
Keywords: Head and Neck Cancer; upper aero digestive tract cancer; Covid19; patient care
MeSH Terms: conditions — Head and Neck Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since its emergence in late December 2019, the SARS-CoV-2 coronavirus has spread rapidly, causing a global health crisis. The disease caused by this highly contagious respiratory virus is called COVID-19. At the beginning of August 2020, there were more than 194,000 confirmed cases in France - including approximately 16,000 cases in the Hauts-de-France area - and more than 30,300 deaths.

Cancer patients are generally susceptible to respiratory infections, and CoV-2-SARS is no exception. Early Chinese studies reported a higher rate of CoV-2-SARS infection in people with cancer (or a history of cancer) than in the general population, with more severe forms and with an increased risk if surgery or chemotherapy is performed in the month prior to infection. The purpose of this study is to describe the management modalities of patients with H&N (Head and Neck) cancer during the COVID-19 pandemic in the Maxillofacial Surgery Department of CHU Amiens-Picardie.

ELIGIBILITY:
Inclusion Criteria:

* patient diagnosed with cancer of the upper aero digestive tract
* patient benefiting from a medical consultation
* patient benefiting from a multidisciplinary consultation meeting for treatment decision between 01/03/2020 and 28/02/2021.

Exclusion Criteria:

* patient diagnosed with cancer other than upper aero digestive tract cancer
* patient whose treatment decision was made before 01/03/2020 (date considered as the beginning of the epidemic at the CHU Amiens-Picardie).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing maxillofacial surgery at the Amiens-Picardie University Hospital between March the 1st 2020 and February the 28th 2021, and in particular from those who have benefited from a multidisciplinary consultation meeting in H&N oncology for treatment decisions during this period.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Variation of delay (in days) between the first cancer consultation and the beginning of the first line of treatment | 6 months
  Variation of delay (in days) between the first cancer consultation and the beginning of the first line of treatment for patients with H&N cancer during the COVID-19 pandemic in the Maxillofacial Surgery Department of CHU Amiens-Picardie.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No